CLINICAL TRIAL: NCT00391690
Title: Evaluation of Bone Markers as Diagnostic Tools for Early Detection of Bone Metastases in Patients With High Risk Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GDE22
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: Serum bone marker; Prostate cancer; Bisphosphonates; Early detection of metastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid — In case of bone metastases: Zoledronic acid every 4 weeks for 3 months.

SUMMARY:
It is the aim of this prospective, single-group, clinical study to assess whether bone parameters can be used as diagnostic tools for early detection of bone metastases in patients with high risk prostate cancer. The usefulness in monitoring zoledronic acid therapy in patients who have developed bone metastases will also be assessed.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically confirmed diagnosis of prostate cancer who have not yet developed bone metastases
* Prostate cancer patients with a rise in PSA under hormone therapy.

PSA criteria:

* Patients who have undergone prostatectomy: any rise in PSA or
* Patients without prostatectomy: 2 consecutive rises in PSA levels relative to a previous reference value, separated by one month. The first measurement must occur one month after the reference value and must be above the reference value. The second confirmatory measurement taken one month after the first measurement must be greater than the first measurement.
* Previous chemotherapy or radiotherapy must have been performed ≥ 8 weeks prior to study entry.
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2 (patients that spend less than 50% of time in bed during the day)
* Adequate liver function - serum total bilirubin concentration less than 1.5 x upper limit of normal value
* Age: ≥ 18 years
* Patient has given written informed consent prior to any study-specific procedures. Patients with psychiatric or addictive disorders which prevent them from giving their informed consent must not enter the study.

Exclusion criteria:

* Prior treatment with a bisphosphonate
* Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute.
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or ≥ 12.0 mg/dl (3.00 mmol/L).
* Patients with clinically symptomatic brain metastases
* History of diseases with influence on bone metabolism such as Paget's disease and primary hyperparathyroidism
* Severe physical or psychological concomitant diseases that might impair compliance with the provisions of the study protocol or that might impair the assessment of drug or patient safety, e.g. clinically significant ascites, cardiac failure, NYHA III or IV, clinically relevant pathologic findings in ECG
* Known hypersensitivity to zoledronic acid or other bisphosphonates
* Use of other investigational drugs 30 days prior to the date of randomization
* Known history or present abuse of alcohol or drugs
* Subjects who, in the opinion of the investigator, are unlikely to cooperate fully during the study
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
• To assess the relationship between change in bone parameters and bone scan with respect to bone metastases | Every 3 months

SECONDARY OUTCOMES:
Assessment of course of bone parameters (PINP, amino-terminal propeptide of procollagen type 1) and (ICTP, Pyridinoline cross-linked carboxyterminal telopeptide of type I collagen) | Every 3 months
Assessment of course of Prostate-specific antigen (PSA) | Every 3 months
Assessment of correlation of bone parameters and PSA | Every 3 months
Assessment of optimal intervals for bone scans based on serum markers | Every 3 months
Assessment of time to rise in bone markers PINP and ICTP | Every 3 months
• Time to detection of bone metastases in bone scan | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Tübingen, Germany

REFERENCES:
- [Result] Lein M, Miller K, Wirth M, Weissbach L, May C, Schmidt K, Haus U, Schrader M, Jung K. Bone turnover markers as predictive tools for skeletal complications in men with metastatic prostate cancer treated with zoledronic acid. Prostate. 2009 May 1;69(6):624-32. doi: 10.1002/pros.20917. PMID 19143027